CLINICAL TRIAL: NCT03324477
Title: Cardiometrically Evaluated NaCl 3% Coload Versus Preload for TURP. A Randomized Controlled Trial.
Brief Title: The Hemodynamic Effects of Hypertonic Saline Preload Versus Coload Measured by Non-invasive Cardiometry in Patients Undergoing TURP Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nazmy Edward Seif (Other)
Responsible Party: Sponsor-Investigator, Nazmy Edward Seif, Clinical Professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 11-2017
Record Dates: First submitted 2017-10-22; First posted 2017-10-27 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Transurethral Resection of Prostate Syndrome
MeSH Terms: interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preload group (Experimental): Patients will receive 4 ml/kg of hypertonic saline 3% via G14 cannula over 15-20 min before the induction of spinal anaesthesia.
  Interventions: Drug: hypertonic saline 3%
- coload group (Experimental): Patients will receive 4 ml/kg of hypertonic saline 3% via G14cannula at the maximal possible rate at the time of identification of C.S.F .
  Interventions: Drug: hypertonic saline 3%

INTERVENTIONS:
Drug: hypertonic saline 3% — hypertonic saline 3% is a type of crystalloid solutions with osmolarity higher than that of plasma
  Other Names: hypertonic saline

SUMMARY:
This study is designed to investigate the relevance of the timing of hypertonic saline administration either as a preload or as a coload on hemodynamic parameters in patients undergoing TURP surgeries.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia is common in elderly males, and this group of patients is commonly associated with different comorbidities especially of the cardiovascular system , this make them at risk of many intraoperative complications. The associated adverse effects arising in both the cardiovascular and nervous systems are known as transurethral resection (TUR) syndrome.Therefore TURP patients need meticulous monitoring of hemodynamics and fluid therapy.

This study is designed to investigate the relevance of the timing of hypertonic saline administration either as a preload or as a coload on hemodynamic parameters in patients undergoing TURP surgeries.

100 ASA physical status I-III male patients scheduled to electively undergo transurethral resection of the prostate under spinal subarachnoid block were included in this study

Preload group (Group P):

50 Patients will receive 4 ml/kg of hypertonic saline (NaCL3%) via G14 cannula over 15-20 min before the induction of spinal anaesthesia.

Co-load group (Group C):

50 Patients will receive 4 ml/kg of hypertonic saline (NaCL3%) via G14 cannula at the maximal possible rate at the time of identification of C.S.F .

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I - III.

Exclusion Criteria:

* Patient refusal.
* Patient in whom spinal anesthesia is absolutely contraindicated.
* Known sensitivity to local anesthetics.
* Preoperative electrolyte imbalance.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
systolic blood pressure | two hours
  systolic blood pressure is measured by mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Nazmy E Seif, MD, Principal Investigator — Cairo University; Manal M Elgohary, MD, Principal Investigator — Cairo University; Manar M Elkholy, MD, Principal Investigator — Cairo University
Locations (1):
- Faculty of Medicine, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided